CLINICAL TRIAL: NCT06920537
Title: Postpartum Cardio-obstetric Rehabilitation After Hypertensive Pregnancy
Brief Title: Postpartum CO Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Mariane Bertagnolli, Assistant Professor, Scientist, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-32-2025-2963
Record Dates: First submitted 2025-03-14; First posted 2025-04-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Gestational Hypertension; Preeclampsia (PE)
Keywords: postpartum rehabilitation; physical exercise; blood pressure; Pelvic Floor; gestational hypertension; pre-eclampsia; small vessels; endothelial function
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research team that will evaluate the participants will be blind to the group - intervention or control (conventional care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rehabilitation Group (Experimental): The rehabilitation Group will be submitted to an 8-week exercise and education program with a hybrid format, delivered by a professional physiotherapist at the Centre Jean-Jacques Gauthier (CJJG). Briefly, one in-person session (60 minutes of aerobic exercise and full-body strength exercise), one online session (30-35 minutes - focus on pelvic floor muscle training, core/abdominals, balance, and stretching exercises), and one pre-recorded video (30 minutes - exercise instructions) will be delivered per week. Participants will use Fitbit Charge-6 to progressively reach daily 10,000 steps throughout the intervention period. Four online educational workshops on healthy lifestyle will be delivered.
  Interventions: Other: Postpartum Cardio-obstetric Rehabilitation Program
- Control group (No Intervention): Control group participants will received the usual care, together with information about the guidelines for physical activity practice, nutritional and risk factor monitoring instructions, pelvic floor exercise instructions, and recommendations to progressively reach daily 10,000 steps according to guidelines . Participants will also receive a Fitbit device.

INTERVENTIONS:
Other: Postpartum Cardio-obstetric Rehabilitation Program — The intervention consists of an 8-week exercise and education program with a hybrid format (in person, virtual and pre-recorded sessions). The aerobic exercise intensity will progressively increase from 50 to 85% of Targeted Heart Rate Range (THRR), calculated for middle-aged women using the maximal heart rate (HR) estimated as 206 - (0.88 x age) . First and second weeks training will target an intensity of 50-65% THRR, third and fourth weeks will target 65 to 75% of THRR, fifth to seventh weeks will target 75 to 80%, and eighth week will target 85%. Participants will use Fitbit Charge-6 to monitor THRR during exercise sessions. Pelvic floor, body alignment/core stability, balance, and low back pain prevention exercises will be added to each in-person session and repeated during the online session. Participants from the intervention group will receive recommendations to progressively reach daily 10,000 steps throughout the intervention period.
  Arms: Rehabilitation Group

SUMMARY:
Some women who develop high blood pressure during pregnancy, such as gestational hypertension or preeclampsia, may continue to have slightly or moderately high blood pressure after giving birth. This can increase their risk of heart disease later in life. Managing blood pressure and adopting a healthy lifestyle after pregnancy could help lower this risk.

Right now, the investigators don't know much about how postpartum rehabilitation programs focused on heart and pregnancy-related health could help women with these conditions. However, a feasibility study suggests that exercise programs might help reduce blood pressure and encourage healthier lifestyles in these women.

In this study, the investigators are testing an 8-week exercise program to see how it affects blood pressure, fitness, and blood vessel health. The investigators will compare the results with a group of women who receive usual healthcare, which includes verbal advice on healthy living but no supervised exercise sessions.

This type of program, called cardio-obstetric rehabilitation, combines exercises for heart health with specialized care for women's health.

DETAILED DESCRIPTION:
Women with severe hypertensive disorders during pregnancy, such as preeclampsia (PE), have a higher risk of heart disease and stroke within five to 10 years of their pregnancy. Because their blood pressure (BP) drops in the postpartum period in comparison to the values they had during pregnancy, the hypertensive disorder can be considered resolved. However, recent studies have shown that their postpartum BP may be higher than before pregnancy. Hypertensive pregnancy has been associated with endothelial and microvascular dysfunction and capillary rarefaction, which could be the key mechanism leading to elevated BP in the postpartum period. Studies have shown that physical exercise promotes BP reduction, stimulates angiogenesis and improves microcirculation in healthy subjects, but also in patients with cardiovascular and metabolic diseases. Therefore, interventions to better monitor BP combined with a healthy lifestyle could help reduce the risk of heart disease in later years. The effects of postpartum cardio-obstetric rehabilitation in women with gestational hypertension (GH) or PE are still unknown. It is of interest to determine whether a postpartum cardio-obstetric rehabilitation program could reduce BP, identifying the possible mechanisms, and stimulate the adoption of a healthy lifestyle with potential long-term health benefits for women.

The main objective of this study is to describe the effects of an 8-week rehabilitation program combining aerobic exercise with obstetric rehabilitation starting between 3 to 6 months postpartum on BP changes, vascular structure and physical activity levels, which could lead to long term health benefits compared to usual care in women with previous GH and PE. The 8-week rehabilitation program will include cardiac (aerobic exercise) and obstetric (pelvic floor training, core and balance) exercises, as well as online education courses about healthy lifestyle. The outcomes will be compared with participants submitted to the usual care in the postpartum. At the end of the study participation period, participants of the control group will be offered to participate in the intervention program (crossing study).

The following outcomes will be evaluated, before and immediately after the intervention: ambulatory and 24-hour BP, arterial stiffness, pulse wave velocity, static retinal vessels analysis, body composition (including body mass index), physical capacity (6-minute walk test), physical activity level (number of daily steps), lipid and glucose profiles, quality of life (SF-36), as well as plasmatic angiogenic biomarkers and the angiogenic function of circulating endothelial cells. Moreover, 6-months post-intervention, participants will be submitted again only to physical evaluation to assess the long-term effects of the intervention program.

Cardio-obstetric rehabilitation is a new field, lacking the description and evaluation of effective programs. The investigators expect that the results obtained from this study will contribute to the design of a patient-oriented rehabilitation program. Our findings will provide the first evidence to support postpartum rehabilitation services in clinics which in turn could lead to long term health benefits to women.

ELIGIBILITY:
Inclusion Criteria:

* are 3 to 6 months postpartum, willing, and able to give informed consent for participation;
* are more than 18 years old;
* are able to access and use a computer, mobile phone and internet (for online sessions);
* were diagnosed with GH (BP higher than 139/89 mmHg after 20 gestational weeks) or PE (BP higher than 139/89 mmHg and proteinuria after 20 gestational weeks) during pregnancy.

Exclusion Criteria:

* have chronic (pre-existing) hypertension (BP>139/89 mmHg pre-pregnancy, <20 weeks' gestation or after 6 weeks postpartum);
* received antihypertensive drug therapy prior to pregnancy or after 6 weeks postpartum;
* are taking beta-blockers for any reason;
* participated in exercise activity programs regularly before 3-month postpartum (more than 2 hour of moderate-to-vigorous exercise per week);
* have any musculoskeletal injury that can limit or contraindicate the practice of exercise;
* have any major contraindications to exercise such as cardiomyopathy, cardiac arrhythmias and conduction abnormalities or congenital heart disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Office Blood Pressure | Baseline, immediately post-intervention, and 6-month post-intervention
  Resting office BP will be measured with the patient in the sitting position after 5 minutes at rest using a validated automated sphygmomanometer according to established practice guidelines . Three readings will be taken at intervals of 2 minutes.
24-hour Ambulatory Blood Pressure | Baseline, immediately post-intervention, and 6-month post-intervention
  24-hour Ambulatory Blood Pressure using OSCAR 2 equipment.

SECONDARY OUTCOMES:
Static Retinal Vascular Analysis | Baseline, immediately post-intervention, and 6-month post-intervention
  Retinal microvasculature imaging will be taken using Static Vessel Analyzer (SVA-T, Imedos) through non-invasive procedures described by Hanssen's team .
Peripheral artery stiffness - PWV | Baseline, immediately post-intervention, and 6-month post-intervention
  Peripheral artery stiffness will be measured using SphygmoCor XCEL system through pulse wave velocity (PWV) as described by Daskalopoulou's team.
Peripheral artery stiffness - PWA | Baseline, immediately post-intervention, and 6-month post-intervention
  The Sphygmocor XCEL system will be used to assess arterial stiffness through Pulse Wave Analysis (PWA), according to the instruction guidelines.
Physical capacity (6MWT) | Baseline, immediately post-intervention, and 6-month post-intervention
  Six-minute walk test will be performed following the protocol described by the American Thoracic Society.
Physical activity levels | Baseline, immediately post-intervention, and 6-month post-intervention
  All participants will receive a wrist worn heart rate and accelerometer monitor (Fitbit Charge 6). This device will be used to monitor physical activity levels (total steps per week) and targeted heart rates during exercise training.
Body composition | Baseline, immediately post-intervention, and 6-month post-intervention
  Body composition will be measure using a bioimpedance scale InBody 570.
Timed Up and Go (TUG) | Baseline, immediately post-intervention, and 6-month post-intervention
  TUG test: The objective of TUG test is to assess mobility, balance and fall-risk. It consists of the participant stand-up from a chair, walk 3 meters, turn, walk back and sit down again. Interpretation: test performed ≤10 seconds indicates normal mobility.
Handgrip strength | Baseline, immediately post-intervention, and 6-month post-intervention
  The maximal handgrip strength will be performed using a manual Jamar Hydraulic Hand Dynamometer.
Glucose | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure glucose at the Biochemistry laboratory of the MUHC.
Angiogenic and proliferative function of peripheral blood ECFCs | Baseline, immediately post-intervention, and 6-month post-intervention
  Endothelial cell function will be assessed by the procedures described by Bertagnolli's team . ECFCs = Endothelial colony forming cell
Plasmatic levels of angiogenic factors - VEGF | Baseline, immediately post-intervention, and 6-month post-intervention
  Serum concentration of angiogenic factors by ELISA following manufacturer instructions - Vascular endothelial growth factor (VEGF)
Heart rate variability | Baseline, immediately post-intervention, and 6-month post-intervention
  R-R intervals will be recorded using a Vantage V2 Polar heart rate monitor at a sampling rate of 1,000 Hz. HRV will be recorded during deep breathing maneuver (continuous cycles) for 4 min in a supine position. HRV will be analyzed using Kubios HRV software following guidelines from the Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology.
Circulating Endothelial Cells (cEC) Function | Baseline, immediately post-intervention, and 6-month post-intervention
  cEC tube formation capacity on matrigel, proliferation, and migration capacities.
Total cholesterol | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure total cholesterol at the Biochemistry laboratory of the MUHC.
Insuline | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure total cholesterol at the Biochemistry laboratory of the MUHC.
Glycated hemoglobin (HbA1c) | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure HbA1c at the Biochemistry laboratory of the MUHC.
LDL cholesterol | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure LDL-cholesterol at the Biochemistry laboratory of the MUHC.
HDL cholesterol | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure HDL cholesterol at the Biochemistry laboratory of the MUHC.
Triglycerides | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure triglycerides at the Biochemistry laboratory of the MUHC.
Brain Natriuretic Peptide (NT-PRO-BNP) | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure NT-PRO-BNP at the Biochemistry laboratory of the MUHC.
C-reactive protein (CRP) | Baseline, immediately post-intervention, and 6-month post-intervention
  Blood draw by venipuncture will be collected to measure C-reactive protein (CRP) at the Biochemistry laboratory of the MUHC.
Plasmatic levels of angiogenic factors - NO | Baseline, immediately post-intervention, and 6-month post-intervention
  Serum concentration of angiogenic factors by ELISA following manufacturer instructions - Nitric Oxide (NO).

OTHER OUTCOMES:
SF-36 Quality of Life Questionnaire (SF-36). | Baseline, immediately post-intervention, and 6-month post-intervention
  Health status will be evaluated based on: SF-36 Quality of Life Questionnaire (SF-36).
Patient Health Questionnaire-9 (PHQ-9) | Baseline, immediately post-intervention, and 6-month post-intervention
  Health status will be evaluated based on: Patient Health Questionnaire-9 (PHQ-9) for depression symptoms
Edinburgh Postnatal Depression Scale (EPDS). | Baseline, immediately post-intervention, and 6-month post-intervention
  Health status will be evaluated based on: Edinburgh Postnatal Depression Scale (EPDS).
Pittsburgh Sleep Quality Index (PSQI). | Baseline, immediately post-intervention, and 6-month post-intervention
  Health status will be evaluated based on: Pittsburgh Sleep Quality Index (PSQI).
Pregnancy Physical Activity Questionnaire (PPAQ). | Baseline, immediately post-intervention, and 6-month post-intervention
  Physical activity will be also evaluated based on Pregnancy Physical Activity Questionnaire (PPAQ).
Duke Activity Status Index (DASI) | Baseline, immediately post-intervention, and 6-month post-intervention
  Physical activity will be also evaluated based on Duke Activity Status Index (DASI)
International Physical Activity Questionnaire (IPAQ). | Baseline, immediately post-intervention, and 6-month post-intervention
  Physical activity will be also evaluated based on International Physical Activity Questionnaire (IPAQ).
Pelvic Floor Distress Inventory (PFDI-20) | Baseline, immediately post-intervention, and 6-month post-intervention
  Pelvic health will be evaluated by Pelvic Floor Distress Inventory (PFDI-20)
Urogenital Distress Inventory (UDI) | Baseline, immediately post-intervention, and 6-month post-intervention
  Pelvic health will be evaluated by Urogenital Distress Inventory (UDI).
Pelvic Floor Impact Questionnaire (PFIQ-7). | Baseline, immediately post-intervention, and 6-month post-intervention
  Pelvic health will be evaluated by Pelvic Floor Impact Questionnaire (PFIQ-7).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital du Sacre-Coer de Montréal - CIUSSS du Nord-de-l'Île-de-Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visser VS, Hermes W, Franx A, Koopmans CM, van Pampus MG, Mol BW, de Groot CJ. High blood pressure six weeks postpartum after hypertensive pregnancy disorders at term is associated with chronic hypertension. Pregnancy Hypertens. 2013 Oct;3(4):242-7. doi: 10.1016/j.preghy.2013.07.002. Epub 2013 Aug 9. PMID 26103803
- [Background] Phan K, Schiller I, Dendukuri N, Gomez YH, Gorgui J, El-Messidi A, Gagnon R, Daskalopoulou SS. A longitudinal analysis of arterial stiffness and wave reflection in preeclampsia: Identification of changepoints. Metabolism. 2021 Jul;120:154794. doi: 10.1016/j.metabol.2021.154794. Epub 2021 May 8. PMID 33971204
- [Background] Magee LA, Pels A, Helewa M, Rey E, von Dadelszen P; Canadian Hypertensive Disorders of Pregnancy (HDP) Working Group. Diagnosis, evaluation, and management of the hypertensive disorders of pregnancy. Pregnancy Hypertens. 2014 Apr;4(2):105-45. doi: 10.1016/j.preghy.2014.01.003. Epub 2014 Feb 25. PMID 26104418
- [Background] Lampinen KH, Ronnback M, Kaaja RJ, Groop PH. Impaired vascular dilatation in women with a history of pre-eclampsia. J Hypertens. 2006 Apr;24(4):751-6. doi: 10.1097/01.hjh.0000217859.27864.19. PMID 16531805
- [Background] Davenport MH, Ruchat SM, Mottola MF, Davies GA, Poitras VJ, Gray CE, Garcia AJ, Barrowman N, Adamo KB, Duggan M, Barakat R, Chilibeck P, Fleming K, Forte M, Korolnek J, Nagpal T, Slater LG, Stirling D, Zehr L. 2019 Canadian Guideline for Physical Activity Throughout Pregnancy: Methodology. J Obstet Gynaecol Can. 2018 Nov;40(11):1468-1483. doi: 10.1016/j.jogc.2018.09.004. Epub 2018 Oct 18. No abstract available. PMID 30343979
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams DJ. Pre-eclampsia and risk of cardiovascular disease and cancer in later life: systematic review and meta-analysis. BMJ. 2007 Nov 10;335(7627):974. doi: 10.1136/bmj.39335.385301.BE. Epub 2007 Nov 1. PMID 17975258
- [Background] Bertagnolli M, Nuyt AM, Thebaud B, Luu TM. Endothelial Progenitor Cells as Prognostic Markers of Preterm Birth-Associated Complications. Stem Cells Transl Med. 2017 Jan;6(1):7-13. doi: 10.5966/sctm.2016-0085. Epub 2016 Jul 27. PMID 28170188